CLINICAL TRIAL: NCT06718777
Title: Effect of Two Different Solutions Used in Pressure Injury Care on Wound Healing Process
Brief Title: Effect of Two Different Solutions on Wound Healing in Pressure Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mensure Turan (Other)
Responsible Party: Sponsor-Investigator, Mensure Turan, Asistant Professor, Şırnak Üniversitesi
Organization: Şırnak Üniversitesi (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/39
Record Dates: First submitted 2024-11-04; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Pressure Injuries; Wound Care; Wound Cleansing
Keywords: pressure injury; %0.1 poliheksanit solution; %0.9 sodium chloride
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.1% polyhexanide (Experimental): 0.1% polyhexanide solution was applied 3 times at 48-hour intervals for pressure ulcer care.
  Interventions: Other: 0.1% polyhexanide Care
- 0.9% NaCl (Experimental): 0.9% sodium chloride solution was applied three times at 48-hour intervals for pressure ulcer care.
  Interventions: Other: 0.9 % NaCl Care

INTERVENTIONS:
Other: 0.1% polyhexanide Care — After the patient was randomized for pressure ulcer care, data were recorded at the first follow-up before care and pressure ulcer care was performed with 0.1% polyhexanide solution. Then, 2 treatments were performed at 48-hour intervals and PUSH scores were recorded before each care. A total of three pressure ulcer care and four follow-ups were performed.
  Arms: 0.1% polyhexanide
Other: 0.9 % NaCl Care — After the patient was randomized for pressure ulcer care, data were recorded at the first follow-up before care and pressure ulcer care was performed with 0.9% sodium chloride. Then, 2 care sessions were performed at 48-hour intervals and PUSH scores were recorded before each care. A total of three pressure ulcer care sessions and four follow-ups were performed.
  Arms: 0.9% NaCl

SUMMARY:
Pressure injuries are a condition that reduces patients' quality of life, increases hospitalization time and healthcare costs. When accompanied by infection and complications, mortality increases. The primary goal in pressure injuries is to prevent their occurrence, but once the injury has occurred, it is to provide effective and appropriate care. It is known that 0.9% sodium chloride (NaCl) is used routinely in pressure ulcer care. In addition, if the effectiveness of 0.1% polyhexanide in pressure ulcer care is demonstrated, it may provide data for its use in wound care. For this purpose, the study was completed as a randomized controlled trial with 32 individuals in the 0.1% polyhexanide group and 31 individuals in the 0.9% NaCl group, totaling 63 individuals.

DETAILED DESCRIPTION:
The European Pressure Ulcer Advisory Panel (EPUAP) and the National Pressure Ulcer Advisory Panel (NPUAP) defined pressure injury (PI) as "Local skin and/or subcutaneous tissue damage caused by pressure alone, or by a combination of pressure and shear, most often occurring over bony prominences". It has been stated that the prevalence of pressure ulcers varies between 0-72.5%, and that it is a condition that reduces the quality of life of patients, increases the length of hospital stay and health care costs. In particular, the accompanying infection and complications of PI cause increased mortality. The primary purpose of PIs is to prevent their occurrence and after the injury occurs, it is necessary to provide care with effective and appropriate methods. The determined method should have the feature that can contribute to wound healing. There are many products and methods with appropriate features that can be used in PIs. In addition to the wet-dry gauze dressing used in wound care from past to present, different care solutions are also used. 0.9% NaCl solutions are frequently used in wound care. Since 0.1% polyhexanide solution is also an effective antiseptic, we thought that its use in PI care would contribute to treatment management by determining its effect on wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who have developed pressure injuries
* Patients who have received informed consent from themselves or their guardians

Exclusion Criteria:

* Patients with clotting problems
* Patients using corticosteroids
* Patients receiving additional medical treatment for wound care

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
PUSH score | From 0th hour to 144th hour
  This scale, developed by NPUAP to evaluate the healing process of pressure injuries, was used in the study to evaluate the healing status of pressure injuries in patients receiving pressure injury care. The pressure injury healing status was monitored with the evaluation criteria in the scale. The lowest score to be received from PUSH is 0, and the highest score is 17. A decrease in the score indicates that the pressure injury has healed.

SECONDARY OUTCOMES:
NPUAP Pressure Sore Classification System | 0th hour
  Staging of pressure ulcers is important to assess the stage of the wound after it has formed to determine effective treatment methods. Staging indicates the severity of the pressure ulcer, its depth, the extent of skin affected, and the extent of tissue damage. The latest update was published by the NPUAP and EPUAP in 2009 as six stages.

CONTACTS AND LOCATIONS:
Overall Officials: Mensure Turan, PhD, Principal Investigator — Şırnak Üniversitesi
Locations (1):
- Gazi Yaşargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No